CLINICAL TRIAL: NCT04706715
Title: ImmunoPET Imaging With 89Zr-DFO-REGN3767 in Patients With Advanced Solid Cancer Prior to and During Treatment With Cemiplimab With or Without Platinum-based Chemotherapy
Brief Title: LAG3 PET Imaging in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202000570
Record Dates: First submitted 2020-12-03; First posted 2021-01-13 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Solid Tumor
Keywords: cancer; immune checkpoint inhibitor; positron emission tomography; LAG-3
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose finding cohort (Experimental): In part A of this imaging trial, a dose finding study will be performed to establish safety, to assess the appropriate protein dose for PET-scanning and to assess the appropriate PET scanning interval. After completion of imaging, patients will start treatment with cemiplimab with or without platinum-based chemotherapy.
  Interventions: Other: 89Zr-DFO-REGN3767; Drug: Cemiplimab
- Feasibility cohort (Experimental): The purpose of part B of the study is to analyze the PK of 89Zr-DFO-REGN3767 in patients before and during treatment with cemiplimab with or without platinum-based chemotherapy.
  Interventions: Other: 89Zr-DFO-REGN3767; Drug: Cemiplimab

INTERVENTIONS:
Other: 89Zr-DFO-REGN3767 — Anti-LAG-3 PET imaging tracer
Drug: Cemiplimab — Cemiplimab 350 mg every 3 weeks with or without platinum-based chemotherapy.

SUMMARY:
This is an investigator-initiated, single-center, open-label clinical trial designed to evaluate the safety and PK of the PET tracer 89Zr-DFO-REGN3767 in patients prior to and during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing informed consent.
2. Patients with histologically confirmed diagnosis of locally advanced or metastatic solid cancer types who, according to the opinion of the investigator, based on available clinical data, may benefit from PD1 antibody with or without platinum-based chemotherapy.
3. At least 1 lesion that is accessible per investigator's assessment and eligible for biopsy according to standard clinical care procedures.
4. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions except for lesions that have progressed after radiotherapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥ 12 weeks.
7. Adequate organ and bone marrow function as defined below:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count ≥1.5 x 109/L
   3. Absolute lymphocyte count ≥0.75 x 109/L
   4. Platelet count ≥100 x 109/L
   5. Serum creatinine ≤1.5 x upper limit of normal (ULN) or estimated glomerular filtration rate > 30 mL/min/1.73 m2. A 24-hour urine creatinine collection may substitute for the calculated creatinine clearance to meet eligibility criteria.
   6. Adequate hepatic function:

   i. Total bilirubin ≤1.5 x ULN (≤3 x ULN if liver tumor involvement); Patients with Gilbert's syndrome do not need to meet total bilirubin requirements, provided their total bilirubin is unchanged from their baseline. Gilbert's syndrome must be documented appropriately as past medical history.

   ii. Aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 x ULN if liver tumor involvement) iii. Alanine aminotransferase (ALT) ≤2.5 x ULN (≤5 x ULN if liver tumor involvement) iv. Alkaline phosphatase (ALP) ≤2.5 x ULN (≤5 x ULN if liver or bone tumor involvement)
8. Signed informed consent.
9. Willingness and ability to comply with all protocol required procedures.

Exclusion Criteria:

1. Treatment with any approved anti-cancer therapy, investigational agent, or participation in another clinical trial with therapeutic intent within 28 days prior to 89Zr-DFO-REGN3767 injection.
2. Prior ICI treatment, including but not limited to anti-PD1 and anti-PD-L1 therapeutic antibodies.
3. Encephalitis, meningitis or uncontrolled seizures in the year prior to inclusion.
4. Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
5. Symptomatic, untreated brain metastasis, leptomeningeal disease, or spinal cord compression. Patients are eligible if central nervous system (CNS) metastases are adequately treated and neurologically stable for at least 2 weeks prior to enrollment.
6. Documented allergic or acute hypersensitivity reaction attributed to antibody treatments.
7. Major surgical procedure other than for diagnosis within 28 days prior to 89Zr-DFO-REGN3767 injection or anticipation of need for a major surgical procedure during the course of the study.
8. For patients that will be treated with cemiplimab in combination with platinum containing chemotherapy, the following additional criteria apply:

   * Age > 70 years
   * Leucopenia <3 x 109/L
   * Estimated glomerular filtration rate < 60 mL/min/1.73 m2
   * Cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), unstable angina, unstable cardiac arrhythmias, myocardial infarction < 3 months ago, or cerebrovascular accident < 6 months ago.
   * Hearing loss
   * Any other exclusion criteria, according to the local clinical practice guidelines for the chosen chemotherapy regimen.
9. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis.

   * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for his study.
   * Patients with controlled type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
10. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.

    • History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
11. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 4 weeks prior to 89Zr-DFO-REGN3767 injection.

    * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g. a one-time of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the sponsor.
    * The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
12. Prior allogeneic bone marrow transplantation or solid organ transplant.
13. Active infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C or tuberculosis infection; or diagnosis of immunodeficiency

    * Patients will be tested for hepatitis C virus (HCV) and hepatitis B virus (HBV) at screening.
    * Patients with known HIV infection who have controlled infection (undetectable viral load (HIV ribonucleic acid (RNA) polymerase chain reaction (PCR)) and CD4 count above 350 either spontaneously or on a stable antiviral regimen are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
    * Patients with hepatitis B who have a controlled infection (serum HBV deoxyribonucleic acid (DNA) PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
    * Patients who are HCV antibody positive who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
    * Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
14. Active infection, that requires systemic antibiotics within 2 weeks prior to 89Zr-DFO-REGN3767 injection.
15. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of 89Zr-DFO-REGN3767, or that may affect the interpretation of the results or render the patient at high risk from complications.
16. Receipt of a live vaccine (including attenuated) within 30 days of planned start of study medication.
17. Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
18. Sponsor employee/member of the clinical site study team and/or his or her immediate family
19. Women with a positive serum chorionic gonadotropin HCG pregnancy test at the screening/baseline visit. Breastfeeding women are also excluded.
20. Women of childbearing potential* and sexually active men who are unwilling to practice highly effective contraception prior to the first dose of study therapy, during the study, and for at least 6 months after the last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Optimal 89Zr-DFO-REGN3767 dose and PET imaging timepoint | 2 years
  Determine the optimal 89Zr-DFO-REGN3767 dose and optimal PET imaging timepoint.
Pharmacokinetics (PK) of 89Zr-DFO-REGN3767 | 2 years
  Description of PK of 89Zr-DFO-REGN3767 by measuring standardized uptake value (SUV) on PET scans performed 0, 2, 4 and/or 7 days after tracer injection.
Incidence of adverse events related to 89Zr-DFO-REGN3767 administration as assessed by CTCAE v5.0 | 2 years
  Safety assessment through summaries of adverse events, changes in laboratory test results (if evaluation is indicated) and changes in vital signs. Adverse event data will be recorded and summarized according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Heterogeneity of 89Zr-DFO-REGN3767 antibody tumor uptake | 2 years
  Heterogeneity of 89Zr-DFO-REGN3767 uptake will be evaluated by measuring standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.
Correlation of tumor tracer uptake with tumor and immune cell LAG3 expression | 2 years
  Results of immunohistochemical (IHC) scoring of immune cell LAG3 expression will be described as a semi-quantitative score using the percentage of positive cells (continuous variable), intensity and pattern of staining (discrete variable). These IHC results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.
Correlation of tumor tracer uptake with response to cemiplimab | 2 years
  Response to therapy with cemiplimab (with or without chemotherapy) will be assessed according to the RECIST or iRECIST guidelines. These results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.
Assessment of changes in tumor and normal organ uptake | 2 years
  Patients enrolled in part B will undergo a PET scan at baseline and another one after 2 treatment cycles. 89Zr-DFO-REGN3767 tracer uptake will be quantified and expressed as standardized uptake value (SUV) in defined volumes of interest (VOIs) for both scans. The results of both PET scans will be compared to assess changes in imaging tracer uptake over time.

CONTACTS AND LOCATIONS:
Overall Officials: E GE de Vries, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groninen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No